CLINICAL TRIAL: NCT06011096
Title: The Effect of Skin-to-Skin Contact and Delayed Cord Clampingon Placental Separation Time, Separation Method, Amount of Postpartum Bleeding and Postpartum Comfort
Brief Title: The Effect of Skin-to-skin Contact on Placental Separation Time, Type, Postpartum Hemorrhage and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahar GÖBEL (Other)
Responsible Party: Sponsor-Investigator, Bahar GÖBEL, Midwife, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Erzurum Atatürk Üniversitesi
Record Dates: First submitted 2023-08-09; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Patient Comfort; Postpartum Hemorrhage; Midwifery; Placenta
Keywords: skin-to-skin contact; placental separation time; Postpartum Comfort; placental separation method; delayed clamping of the umbilical cord; midwife
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group with skin-to-skin contact and delayed cord clamping (Experimental): In this arm, skin-to-skin contact and delayed cord clamping are performed between mother and baby.
  Interventions: Other: skin-to-skin contact and delayed cord clamping
- The group without skin-to-skin contact and early cord clamping (Experimental): In this arm, skin-to-skin contact and delayed cord clamping are not performed between mother and baby.
  Interventions: Other: avoiding skin-to-skin contact and early cord clamping

INTERVENTIONS:
Other: skin-to-skin contact and delayed cord clamping — Placental separation time, separation method, amount of postpartum bleeding and postpartum comfort were evaluated with skin-to-skin contact and late cord clamping after delivery.
  Arms: the group with skin-to-skin contact and delayed cord clamping
Other: avoiding skin-to-skin contact and early cord clamping — After delivery, placental separation time, separation method, amount of postpartum bleeding and postpartum comfort were evaluated without skin-to-skin contact and late cord clamping.
  Arms: The group without skin-to-skin contact and early cord clamping

SUMMARY:
It is aimed to determine the late cord clamping with early skin-to-skin contact in primiparous pregnant women who delivered vaginally, according to placental separation time, separation method, amount of postpartum bleeding and postpartum comfort.

DETAILED DESCRIPTION:
The research is an experimental type randomized controlled trial. The data of the research gathered in the delivery room clinic of Erzurum City Hospital affiliated to the Ministry of Health in Erzurum city center between 02.11.2022 and 10.06.2023. The study was completed with 126 primiparous pregnants, 63 of whom were controls and 63 of whom were experimental, randomized in the clinic. "Personal Information Form" and "Postpartum Comfort Scale" prepared by the researcher were used to collect the data of the study.

control group

* Pregnant women who met the criteria for admission to the delivery room were selected, the institution's routine policies were implemented.
* The mother was informed about the study and written consent was obtained.
* Hospital routine practices continued until birth.
* The stopwatch is started the moment the baby is born.
* After birth, the umbilical cord was clamped immediately without skin-to-skin contact between the mother and the baby, and the baby was taken to routine care.
* Signs of placental separation were monitored with a stopwatch, and it was noted at what minute the symptoms were seen.
* Placental delivery time and separation type were noted in the relevant part of the form.
* According to the routines taken from each hospitalized patient in institutional policies, the volunteer's entry hemoglobin and hematocrit values were noted on the form.
* The Personal Information Form consisting of 22 questions and the Postpartum Comfort scale were administered to the mother at the end of the follow-up period in the delivery room (2 hours later).
* From the 6th hour blood values found in the hospital routine, the mother's hemoglobin and hematocrit values were noted on the form.

Experimental group

* Pregnant women who met the criteria for admission to the delivery room were selected, the institution's routine policies were implemented.
* The mother was informed about the study and written consent was obtained.
* Hospital routine practices continued until birth.
* The stopwatch is started the moment the baby is born.
* The baby was placed on the mother's chest, it was waited for 60-90 seconds in skin-to-skin contact, and breastfeeding was tried. At the end of the period, the umbilical cord was clamped and the baby was placed under a radiant heater and routine care was continued.
* Signs of placental separation were monitored with a stopwatch, and it was noted at what minute the symptoms were seen.
* Placental delivery time and separation type were noted in the relevant part of the form.
* According to the routines taken from each hospitalized patient in institutional policies, the volunteer's entry hemoglobin and hematocrit values were noted on the form.
* During the repair of episiotomy or desuria, if any, in the mother, skin-to-skin contact was made between the baby and the mother for 1 hour without disrupting the procedures.
* The Personal Information Form consisting of 22 questions and the Postpartum Comfort scale were administered to the mother at the end of the follow-up period in the delivery room (2 hours later).
* From the 6th hour blood values found in the hospital routine, the mother's hemoglobin and hematocrit values were noted on the form.

ELIGIBILITY:
Inclusion Criteria:

* for pregnant women

  1. Those who agreed to participate in the research
  2. 18-49 years old
  3. Firstborn (nulliparous)
  4. Have 37-42 weeks of pregnancy
  5. The baby in head presentation
  6. No prenatal risk pregnancy
  7. No risk during and after birth
* for newborns

  1. Absence of any health problems or congenital diseases,
  2. No need for resuscitation after birth.
  3. APGAR score of 8 points or more

Exclusion Criteria:

1. Births less than 37 weeks
2. Multiparity
3. Any complications in the mother or baby
4. Removal of the placenta by intervention rather than spontaneous separation

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primiparous women giving birth vaginally
Enrollment: 126 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Skin-to-skin contact and delayed cord clamping affect placental separation time. | 0-30 minute
  It shortens the placental separation time in women who have had a vaginal delivery with skin-to-skin contact and delayed clamping of the cord.
Skin-to-skin contact and delayed cord clamping affect the amount of postpartum bleeding. | 0-6 hours
  Skin-to-skin contact and delayed cord clamping reduce the amount of postpartum hemorrhage in women who deliver vaginally.
Skin-to-skin contact and delayed cord clamping have no effect on the type of placental separation. | 0-30 minute
  Determination of the effect of skin-to-skin contact and delayed cord clamping on the type of placental separation.
Skin-to-skin contact and delayed cord clamping affect the level of postpartum comfort. | 2 hours
  Increasing the postpartum comfort level of women who had vaginal delivery with skin-to-skin contact and delayed cord clamping.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Göbel, Principal Investigator — Midwife
Locations (1):
- Erzurum City Hospital, Erzurum, Turkey (Türkiye)